CLINICAL TRIAL: NCT03770858
Title: A Single Arm, Prospective Clinical Study Using Novel Wearable Sensors to Assess the Improvement of Nocturnal Scratch Behavior and Sleep Quality in Children With Mild-to-moderate Atopic Dermatitis Treated With Topical Crisaborole
Brief Title: Wearable Skin Sensors to Assess Nocturnal Scratch Behavior
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Other Study IDs: 052018SX
Record Dates: First submitted 2018-09-06; First posted 2018-12-10 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Atopic Dermatitis
Keywords: Wearables; Atopic Dermatitis; Scratch sensor
MeSH Terms: conditions — Dermatitis, Atopic | interventions — crisaborole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Crisaborole and wearable sensor: Subjects will apply topical crisaborole twice daily to the affected atopic dermatitis areas for three weeks.
  Interventions: Drug: Crisaborole; Device: Scratch sensor

INTERVENTIONS:
Drug: Crisaborole — Subject to apply topical crisaborole twice daily to the affected atopic dermatitis areas
Device: Scratch sensor — advanced, flexible and wearable skin sensor

SUMMARY:
Pilot study of flexible and wearable sensor to monitor nocturnal scratching behavior

DETAILED DESCRIPTION:
Present an advanced flexible, and wearable sensor intimately coupled to the skin that can measure the full spectrum of relevant physiological parameters associated with atopic dermatitis including scratch count, scratch duration, scratch intensity, heart rate, heart rate variability and respiratory rate.

ELIGIBILITY:
Inclusion Criteria:

* Participants with mild to moderate atopic dermatitis ages 2 years or older. This will be determined by clinical diagnosis of AD according to the Hanifin and Rajka criteria with a baseline Investigators Global Assessment score of mild (2) or moderate (3)
* Systemic therapy use (e.g. oral corticosteroid, cyclosporine, methotrexate, phototherapy) within 28 days of subject enrollment
* Topical corticosteroid use or topical calcineurin inhibitor use within 14 days of subject enrollment
* Willingness and ability to set up an infrared video camera nightly
* Willing to apply topical crisaborole twice daily to affected atopic dermatitis areas of the body

Exclusion Criteria:

* Active skin or systemic infection
* Inability to operate a smartphone or video camera
* Active atopic dermatitis on he dorsum of the hand or suprasternal notch

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with mild to moderate atopic dermatitis
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Percent agreement of scratching between the experimental sensor and the infrared camera | 3 weeks

SECONDARY OUTCOMES:
Improvement of sleep parameters (time asleep) measured by the experimental sensor during treatment | 3 weeks
  Baseline compared to treatment time points will be compared in units of time (minutes/hours)
Improvement of sleep parameters (time until onset of sleep) measured by the experimental sensor | 3 weeks
  Baseline compared to treatment time points will be compared in units of time (minutes/hours)
Improvement of sleep parameters (heart rate) measured by the experimental sensor | 3 weeks
  Baseline compared to treatment time points will be compared in units of beats/min
Improvement of sleep parameters (respiratory rate) measured by the experimental sensor | 3 weeks
  Baseline compared to treatment time points will be compared in units of breaths/min.

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Xu, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No